CLINICAL TRIAL: NCT01338688
Title: the Change of the Tetanus Antibody Titer After Single Injection of Tetanus Vaccine and Simultaneous Injection of Tetanus Immunoglobulin With Tetanus Vaccine?
Brief Title: The Change of the Tetanus Antibody Titer After Single Injection of Td and Simultaneous Injection of TIG With Td
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Boramae Hospital (Other)
Responsible Party: Jong Hwan Shin, Seoul National University-Seoul Metropolitan Goverment Boramae Hospital
Other Study IDs: Td-TIG
Record Dates: First submitted 2011-04-07; First posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Tetanus
MeSH Terms: conditions — Tetanus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Td ,Td and TIG

SUMMARY:
The investigators want to determine whether TIG influences the formation of tetanus antibody after simultaneous tetanus vaccination according to age and the time-interval of the last tetanus vaccination.

DETAILED DESCRIPTION:
When an injured patient visits the ED, unnecessary injection of tetanus immunoglobulin (TIG) may cause side effects and also increase the medical expense.5 Further, the opportunity of assessing a rising tetanus antibody titer may be missed after simultaneous injection of tetanus-diphtheria vaccine (Td) and TIG. According to age, the elevation of the tetanus antibody titer after tetanus prophylaxis might be not equivalent because of different levels of basal immunity and the time-interval of the last tetanus vaccination. Therefore, we wanted to determine whether TIG influences the formation of tetanus antibody after simultaneous tetanus vaccination according to age and the time-interval of the last tetanus vaccination.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult volunteers

Exclusion Criteria:

* immunocompromised
* febrile
* allergy to the vaccine constituents
* previous tetanus immunization within 5 years
* medical and non-medical employees

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adult over twenty
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The change from baseline in tetanus antibody titer at 4weeks, 6 months and 12months | Baseline, 4 weeks, 6 months, 12 months
  The tetanus antibody titers were determined by ELISA and the results were reported in IU/mL. The measurement of tetanus antibody titer at 4 weeks should be needed to check the peak titer after vaccination. the change of tetanus antibody titers were calculated by geometric mean titers(GMTs), and we compared the GMTs between the groups(Td vs Td-TIG)at baseline, 4weeks, 6months, and 12 months by independent T-test.

CONTACTS AND LOCATIONS:
Overall Officials: JongHwan Shin, Principal Investigator — Seoul National University Boramae Hospital